CLINICAL TRIAL: NCT05808179
Title: Passive Phototherapy to Improve Sleep in Teens
Brief Title: Shifting Sleep Timing in Teens
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Professor, Stanford University
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HD102344 (NIH)
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Sleep Insufficiency; Sleep; Adolescent Behavior
MeSH Terms: conditions — Sleep Deprivation; Adolescent Behavior | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light + Cognitive Behavioral Therapy (CBT) (Experimental): 1 hour of light flashes (typical wake time - 75 min → typical wake time - 15 min) and cognitive behavioral therapy
  Interventions: Device: Light; Behavioral: CBT
- Sham light + CBT (Active Comparator): 1 hour of sham light flashes (one flash) and cognitive behavioral therapy
  Interventions: Behavioral: CBT; Device: Sham Light

INTERVENTIONS:
Device: Light — Broad-spectrum white light flashes are ~4000 lux, 2 msec long, occur every 20 s
  Arms: Light + Cognitive Behavioral Therapy (CBT)
Behavioral: CBT — Cognitive behavioral therapy including psychoeducation, sleep hygiene, stimulus control, activity scheduling, motivational interviewing
Device: Sham Light — Broad-spectrum white light flashes are ~4000 lux, 2 msec long, occur once
  Arms: Sham light + CBT

SUMMARY:
The goal of this clinical trial is to determine whether a combination of a novel lighting intervention and a behavioral intervention are able to increase total sleep time in adolescents. The main questions this trial aims to answer are whether this combination therapy is able to meaningfully increase total sleep time in adolescents, and do so over a sustained period of time, and whether such a changes is associated with concomitant changes in mood and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-18 and a full-time student in grades 9-12
2. Male or female
3. Willing and with a schedule permitting them to go to bed at an earlier time
4. Planning on sleeping at home in their bedroom for at least 75% of the study

Exclusion Criteria:

1. Currently taking any medications (including over-the-counter medications, e.g., melatonin) specifically for the treatment of sleep disorders
2. Sleep only in the prone (face-down) position

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Total sleep time | 20 weeks
  Average nightly total sleep time

SECONDARY OUTCOMES:
Melatonin timing | 8 weeks
  Timing of the onset of salivary melatonin
Mood | 20 weeks
  Score on the Center for Epidemiologic Studies Depression Scale for Children. Scored 0-60 with higher scores indicating greater depressive symptomatology.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made freely available on Dryad.com. Study protocol, analysis plan, consent form (unsigned), and analytic code will be made available upon request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Keskinel D, Karan M, Kaplan KA, Mirchandaney R, Asarnow L, Zeitzer JM. Piloting a brief digital behavioral intervention for adolescent sleep. Sleep Sci Pract. 2025;9(1):34. doi: 10.1186/s41606-025-00157-4. Epub 2025 Oct 31. PMID 41180604

DOCUMENTS (1):
  • Informed Consent Form (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT05808179/ICF_000.pdf